CLINICAL TRIAL: NCT03037021
Title: Improving Sickle Cell Disease (SCD) Care Using Web-based Guidelines, Nurse Care Managers and Peer Mentors in Primary Care and Emergency Departments in Central North Carolina
Brief Title: Improving Sickle Cell Disease (SCD) Care Using Web-based Guidelines
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00073506; 1U01HL133964-01 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2017-01-31 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2018-08

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Needs Assessment; Barriers to care; Access to care; Primary care
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (4):
- SCD Adult Patients: Focus group or individual interview and survey
- SCD Adolescent Patients: Focus group or individual interview and survey
- SCD Healthcare Providers: Focus group or individual interview and survey
- Parents of SCD Adolescents: Focus group or individual interview and survey

SUMMARY:
The overall goal of this proposed project is to 1) increase co-management between sickle cell specialists and primary care providers (PCP's); 2) increase the use of hydroxyurea (HU) which prevents Vaso-Occlusive Episode (VOE), EDs and subsequent hospitalizations, and death; 3) identify and link patients not receiving primary or SCD specialty care to care, and 4) shift healthcare use from EDs and hospitalizations to primary and specialty co-management. Many persons with SCD experience a poor quality of life, serious medical complications and frequent painful events that require treatment from SCD specialty care, primary care and emergency department (ED) providers. There are two dominating models of care in the United States; neither are ideal. Many people with SCD have all of their healthcare needs addressed by sickle cell specialists who do not typically provide primary care and are often geographically distant from the patients' home. Other sickle cell patients receive all of their care in EDs. Both models are inadequate and result in an alarmingly high number of ED visits for many patients. Current care models are neither cost efficient nor promoting optimal patient outcomes. To improve outcomes, the investigators will implement a new model of care for SCD using nurse care managers, web based-interactive algorithms, and test if additional patient provided coaching can improve outcomes.

DETAILED DESCRIPTION:
To inform the model, the investigators will conduct an initial in-depth multi-level assessment of the barriers to care and implementation of the NHLBI "Evidence-Based Management of Sickle Cell Disease". With barriers and facilitators identified at the patient, provider, healthcare organization and community levels, the investigators will develop another study evaluation interventions that may improve the barriers.

ELIGIBILITY:
Inclusion Criteria:

- SCD patients in the 31 geographic counties surrounding Duke with genotypes Hemoglobin SS, SC, Sβ° or, Sβ+.

and -Parents of 15-20 year old SCD patients in the 31 geographic counties surrounding Duke with genotypes Hemoglobin SS, SC, Sβ° or Sβ+.

and

-Healthcare providers of sickle cell patients in the 31 geographic counties surrounding Duke

Exclusion Criteria:

* Non-English speaking

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population includes 15-45 year olds with and SCD, parents of 15-20 year olds with SCD and healthcare providers of patients with SCD residing in 31 specified counties in Central North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Barriers to primary care as measured by Focus Groups./interviews | 60 Minutes after focus group or interview
  Qualitative analysis will be used to analyze interviews and focus groups.
Barriers to specialty care as measured by Focus Groups./interviews | 60 Minutes after focus group or interview
  Qualitative analysis will be used to analyze interviews and focus groups.
Barriers to ED care as measured by Focus Groups./interviews | 60 Minutes after focus group or interview
  Qualitative analysis will be used to analyze interviews and focus groups.
Barriers to primary care as measured by Survey | Approximately 30-45 minutes
  Descriptive statistics will be used to summarize the survey data.
Barriers to specialty care as measured by Survey | Approximately 30-45 minutes
  Descriptive statistics will be used to summarize the survey data.
Barriers to ED care as measured by Survey | Approximately 30-45 minutes
  Descriptive statistics will be used to summarize the survey data.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States